CLINICAL TRIAL: NCT01704924
Title: Prospective Observation of Wound Healing With Prevena Incision Management System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No study subjects enrolled, Investigator decided to cancel the project
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Gregory R. Evans, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KCI-2011-8268
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Scarring
Keywords: Prevena; negative pressure wound therapy; Incisional wound vac
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena (Active Comparator): Incision with prevena device overlying
  Interventions: Device: Prevena
- Standard of Care dressing (Active Comparator): Prevena device is not used
  Interventions: Procedure: Standard of Care Dressing

INTERVENTIONS:
Device: Prevena — Device will be applied at end of procedure over closed incision
  Arms: Prevena
Procedure: Standard of Care Dressing — Dressing applied as Standard of Care
  Arms: Standard of Care dressing

SUMMARY:
This study aims to assess the quality of wound healing in abdominal scars with and without the Prevena Incision Management System. The hypothesis is that Prevena will lead to improved wound healing with less swelling, bruising, and inflammation, as well as less potential for infection, seroma, and dehiscence.

DETAILED DESCRIPTION:
The quality of wound healing can be of the utmost importance for patients undergoing large abdominal surgery. Incisional negative pressure wound therapy has been observed to decrease seroma and infection rates in high risk patients. This study aims to quantify the effect, if any, that negative pressure wound therapy has on closed incisions. The technology may provide benefits even in lower risk patients.

ELIGIBILITY:
Inclusion Criteria:

* abdominal procedure with incision >20cm
* must be >18 years of age

Exclusion Criteria:

* <18 years of age
* history of allergy or reaction to adhesives
* pregnant or anticipated pregnancy within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Scarring | 0-6 months
  Assess quality of scar: hypertrophy, hyperpigmentation, etc

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Evans, MD, Principal Investigator — The University of California Irvine
Locations (1):
- University of California at Irvine, Orange, California, United States

REFERENCES:
- [Background] Pachowsky M, Gusinde J, Klein A, Lehrl S, Schulz-Drost S, Schlechtweg P, Pauser J, Gelse K, Brem MH. Negative pressure wound therapy to prevent seromas and treat surgical incisions after total hip arthroplasty. Int Orthop. 2012 Apr;36(4):719-22. doi: 10.1007/s00264-011-1321-8. Epub 2011 Jul 15. PMID 21761149
- [Background] Stannard JP, Volgas DA, McGwin G 3rd, Stewart RL, Obremskey W, Moore T, Anglen JO. Incisional negative pressure wound therapy after high-risk lower extremity fractures. J Orthop Trauma. 2012 Jan;26(1):37-42. doi: 10.1097/BOT.0b013e318216b1e5. PMID 21804414
- See also: Prevena Product Website — http://www.kci1.com/KCI1/prevena